CLINICAL TRIAL: NCT03495856
Title: Feasibility of a 4-week, Adapted Mindfulness Program for Adults With Chronic Pain
Brief Title: 4-week Mindfulness Program for Adults With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-2948; 2KR941702 (Other Grant/Funding Number: North Carolina Translational and Clinical Sciences Institute)
Record Dates: First submitted 2018-03-21; First posted 2018-04-12 (Actual); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-03

CONDITIONS: Chronic Pain
Keywords: Mindfulness-based stress reduction; Mindfulness; chronic pain; Feasibility; Intervention
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Single-group, mixed methods repeated measures design (pre and post assessments)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Training For Chronic Pain (Experimental): The intervention is adapted from the mindfulness-based stress reduction program. The adapted mindfulness training program consists of four, weekly 90 minute group sessions that focus on education on chronic pain and mindfulness, instruction and in-class mindfulness skills practice, and group discussion.
  Interventions: Behavioral: Mindfulness Training For Chronic Pain

INTERVENTIONS:
Behavioral: Mindfulness Training For Chronic Pain — 4-week group Mindfulness training program for adults with chronic pain

SUMMARY:
The objective of this study is to determine the feasibility and acceptability of a 4-week mindfulness training program for adults with chronic pain (noncancer related). The intervention is based on the MIndfulness-based Stress Reduction Program, an 8-week mindfulness training program developed to help people manage stress-related and chronic conditions. The adapted mindfulness intervention will consist of four, weekly 1 hour and 30 minute group sessions that are modified from the original program to fit the shorter length and to directly address chronic pain management. Participants will complete pre- and post-intervention surveys and daily mindfulness practice diaries, all online. The surveys will help us determine if participants experience decreased pain interference, increased quality-of-life, and increased psychological well-being over the course of the intervention. Participants will also complete a post-intervention telephone interview to help determine satisfaction with the intervention and areas where the intervention can be improved.

ELIGIBILITY:
Inclusion Criteria:

* One or more chronic noncancer pain diagnoses (daily pain for at least 3 months)
* Has a pain management provider
* Reports more than minimal pain bothersomeness and interference in general activities
* Able to read and understand English

Exclusion Criteria:

* Diagnosis of mental illness with psychotic features
* History of inpatient admission for psychiatric disorder in past 2 years
* Active alcohol or substance abuse within the past year
* Has completed a mindfulness-based stress reduction or other mindfulness course; has or previously had a regular mindfulness meditation practice.
* Unable or unwilling to comply with study procedures (online questionnaires and practice diaries, 4 weekly intervention sessions, home practice, and one semi-structured phone interview).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Brintz, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Brintz CE, Polser G, Coronado RA, French B, Faurot KR, Gaylord SA. Are Formal and Informal Home Mindfulness Practice Quantities Associated With Outcomes? Results From a Pilot Study of a Four-Week Mindfulness Intervention for Chronic Pain Management. Glob Adv Integr Med Health. 2024 Feb 29;13:27536130241236775. doi: 10.1177/27536130241236775. eCollection 2024 Jan-Dec. PMID 38434590

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Dates: April 2018 to September 2018 Recruitment Setting: Medical clinics; University/Medical center campus and email listserve
Groups:
- Mindfulness Training: 4-week mindfulness skills group for adults with chronic pain
Period: Overall Study
Arm/Group | Mindfulness Training
Started | 23
Completed | 22
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis includes all 23 participants who enrolled and completed the baseline assessment.
Arm/Group | Mindfulness Training
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.00 (15.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23
Years with chronic pain [Mean (Standard Deviation); unit: years] | 6.9 (7.2)
Education [Count of Participants; unit: Participants]
  Less than high school | 0
  High School diploma or equivalent | 1
  Some college, no college degree | 5
  College degree or greater | 16
  Unknown | 1
Yearly Household Income [Count of Participants; unit: Participants]
  Less than $20,000 | 5
  $20,000 to 39,999 | 2
  $40,000 to $59,999 | 4
  $60,000 to $79,999 | 2
  $80,000 + | 8
  Unknown | 2
Source/location of pain [Count of Participants; unit: Participants]
  Back | 18
  Arthritis | 11
  Fibromyalgia | 4
  Neck | 12
  Neuropathy | 11
  Headache/migraine | 7
  Pelvic | 4
  Other | 8

OUTCOME MEASURES:

1. Primary Outcome: Feasibility - Study Retention
Description: Proportion of participants enrolled who completed the study
Time Frame: 4 weeks
Population: All participants who enrolled and completed the baseline assessment
Measure: Mean (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Mindfulness Training
Number analyzed (Participants) | 23
Proportion of participants | 0.96 [0.87 to 1.04]

2. Primary Outcome: Feasibility - Session Attendance
Description: Average sessions attended (proportion)
Time Frame: 4 weeks (intervention weeks 1-4)
Measure: Mean (95% Confidence Interval); unit: Proportion of sessions
Arm/Group | Mindfulness Training
Number analyzed (Participants) | 23
Proportion of sessions | 0.77 [0.58 to 0.96]

3. Primary Outcome: Credibility and Expectancy Questionnaire Scores
Description: Credibility and Expectancy Questionnaire. Each item is scored separately and rated on a scale from 1 [not at all] to 10 [very]. Scores for each item range from 1-10, with higher ratings indicating higher credibility and expectancy.
Time Frame: Intervention week 2
Population: Participants who completed the measure after session 2 (week 2)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Training
Number analyzed (Participants) | 22
units on a scale
  How logical is the mindfulness program | 6.4 (2.4)
  Confidence that program will improve chronic pain | 6.0 (2.2)
  Confidence in recommending program to friend | 6.4 (2.8)
  How important we make this available to others | 7.3 (2.7)
  Believe program would decrease other problems? | 7.6 (1.3)

4. Primary Outcome: Acceptability - Intervention Satisfaction
Description: Question assessing participants satisfaction with the intervention
Time Frame: 4 weeks (within one week post-intervention)
Population: Participants who completed the post-assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Training
Number analyzed (Participants) | 22
Participants
  Very dissatisfied | 0
  Moderately dissatisfied | 0
  Slightly dissatisfied | 1
  Neutral | 1
  Slightly satisfied | 1
  Moderately satisfied | 7
  Very satisfied | 12

5. Secondary Outcome: Pain Intensity Scores
Description: Pain intensity rating: 1 item from the Patient Reported Outcomes Measurement Information System (PROMIS), with pain intensity rated on 0-10 scale with lower values indicating less pain, or better outcome.
Time Frame: Baseline and 4 weeks (pre to post-intervention)
Population: Participants who completed baseline and post-assessments
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness Training
Number analyzed (Participants) | 22
units on a scale
  Pre | 5.91 (2.05)
  Post | 5.14 (1.86)
Statistical Analysis 1: Comparison: Mindfulness Training; Test type: Other — within-group paired t-test; p = 0.05, t-test, 2 sided — The a priori threshold for statistical significance was p less than or equal to 0.05. That calculated p-value in the statistical hypothesis test was equal to 0.05; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-1.55 to 0.00], Standard Error of Mean .37

6. Secondary Outcome: Pain Interference Scores
Description: Pain Interference short-form 6b, Patient Reported Outcomes Measurement Information System scale. Raw scores were converted using the HealthMeasures scoring service to standardized T-Scores with M=50, SD=10 and ranging from 20 to 80. A lower score indicates lower pain interference, or a better outcome.
Time Frame: Baseline and 4 weeks (pre to post-intervention)
Population: Participants who completed baseline and post assessments
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Mindfulness Training
Number analyzed (Participants) | 22
T-score
  Pre | 63.76 (7.31)
  Post | 60.10 (5.65)
Statistical Analysis 1: Comparison: Mindfulness Training; Test type: Other — within-group paired t-test; p = 0.017, t-test, 2 sided; Mean Difference (Final Values) = -3.67, 95% CI 2-sided [-6.63 to -0.71], Standard Error of Mean 1.42

7. Secondary Outcome: Physical Functioning Scores
Description: Physical functioning short-form 4a - Patient Reported Outcomes Measurement Information System scale. Raw scores were converted using the HealthMeasures scoring service to standardized T-Scores with M=50, SD=10 and ranging from 20 to 80. A higher score indicates higher physical functioning, or a better outcome.
Time Frame: Baseline and 4 weeks (pre to post-intervention)
Population: Participants who completed baseline and post assessments
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Mindfulness Training
Number analyzed (Participants) | 22
T-score
  Pre | 38.17 (5.35)
  Post | 38.22 (6.81)
Statistical Analysis 1: Comparison: Mindfulness Training; Test type: Other — Within-group paired t-test; p = 0.938, t-test, 2 sided; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-1.39 to 1.50], Standard Error of Mean 0.70

8. Secondary Outcome: Depression Short-Form 4a Scores
Description: Depression short-form 4a - Patient Reported Outcomes Measurement Information System scale. Raw scores were converted using the HealthMeasures scoring service to standardized T-Scores with M=50, SD=10 and ranging from 20 to 80. A lower score indicates less depression, a better outcome.
Time Frame: Baseline and 4 weeks (pre to post-intervention)
Population: Participants who completed baseline and post assessments
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Mindfulness Training
Number analyzed (Participants) | 22
T-score
  Pre | 56.82 (9.75)
  Post | 53.49 (8.62)
Statistical Analysis 1: Comparison: Mindfulness Training; Test type: Other — Within-group paired t-test; p = 0.005, t-test, 2 sided — The a priori threshold for statistical significance was p less than or equal to 0.05; Mean Difference (Final Values) = -3.34, 95% CI 2-sided [-5.53 to -1.15], Standard Error of Mean 1.05

9. Secondary Outcome: Anxiety Short-Form 4a Scores
Description: Anxiety short-form 4a - Patient Reported Outcomes Measurement Information System. Raw scores were converted using the HealthMeasures scoring service to standardized T-Scores with M=50, SD=10 and ranging from 20 to 80. Lower scores represent lower anxiety, a better outcome.
Time Frame: Baseline and 4 weeks (pre to post-intervention)
Population: Participants who completed baseline and post assessments
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Mindfulness Training
Number analyzed (Participants) | 22
T-score
  Pre | 59.06 (9.44)
  Post | 56.84 (8.02)
Statistical Analysis 1: Comparison: Mindfulness Training; Test type: Other — Within-group paired t-test; p = 0.124, t-test, 2 sided; Mean Difference (Final Values) = -2.21, 95% CI 2-sided [-5.09 to 0.66], Standard Error of Mean 1.38

10. Secondary Outcome: Sleep Disturbance Short-Form 4a Scores
Description: Sleep disturbance short-form 4a - Patient Reported Outcomes Measurement Information System. Raw scores were converted using the HealthMeasures scoring service to standardized T-Scores with M=50, SD=10 and ranging from 20 to 80. Lower scores represent less sleep disturbance, a better outcome.
Time Frame: Baseline and 4 weeks (pre to post-intervention)
Population: Participants who completed baseline and post-assessment
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Mindfulness Training
Number analyzed (Participants) | 22
T-score
  Pre | 56.52 (7.79)
  Post | 51.83 (9.75)
Statistical Analysis 1: Comparison: Mindfulness Training; Test type: Other — Within-group paired t-test; p = 0.001, t-test, 2 sided; Mean Difference (Final Values) = -4.69, 95% CI 2-sided [-7.30 to -2.07], Standard Error of Mean 1.26

11. Other Pre Specified Outcome: Perceived Stress Scale Scores
Description: Perceived Stress Scale - 4 item version. Possible scores range from 0-16. Lower scores indicate lower perceived stress, a better outcome.
Time Frame: Baseline and 4 weeks (pre to post-intervention)
Population: Participants who completed baseline and post assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training
Number analyzed (Participants) | 22
score on a scale
  Pre | 7.23 (3.70)
  Post | 5.95 (3.55)
Statistical Analysis 1: Comparison: Mindfulness Training; Test type: Other — Within-group paired t-test; p = 0.018, t-test, 2 sided; Mean Difference (Final Values) = -1.27, 95% CI 2-sided [-2.31 to -0.24], Standard Error of Mean 0.50

12. Other Pre Specified Outcome: Positive Affect and Well-being Scores
Description: Positive Affect and Well-being Scale - 9 items. This scale comes from the Neurological Quality of Life Measurement System (Neuro QOL). Raw scores were converted using the HealthMeasures scoring service to standardized T-Scores with M=50, SD=10 and ranging from 20 to 80. Higher scores indicate greater positive affect and well-being, a better outcome.
Time Frame: Baseline and 4 weeks (pre to post-intervention)
Population: Participants who completed baseline and post assessments
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Mindfulness Training
Number analyzed (Participants) | 22
T-score
  Pre | 47.86 (7.41)
  Post | 50.66 (7.89)
Statistical Analysis 1: Comparison: Mindfulness Training; Test type: Other — Within-group paired t-test; p = 0.016, t-test, 2 sided; Mean Difference (Final Values) = 2.79, 95% CI 2-sided [0.58 to 5.01], Standard Error of Mean 1.07

13. Other Pre Specified Outcome: Pain Catastrophizing Scale Scores
Description: Pain Catastrophizing Scale. Scores range from 0-52, with higher scores indicating more pain catastrophizing, or worse outcome.
Time Frame: Baseline and 4 weeks (pre to post-intervention)
Population: Participants who completed baseline and post assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training
Number analyzed (Participants) | 22
score on a scale
  Pre | 23.64 (12.79)
  Post | 18.68 (12.38)
Statistical Analysis 1: Comparison: Mindfulness Training; Test type: Other — Within-group paired t-test; p = 0.002, t-test, 2 sided; Mean Difference (Final Values) = -4.96, 95% CI 2-sided [-7.88 to -2.03], Standard Error of Mean 1.41

14. Other Pre Specified Outcome: Chronic Pain Acceptance Scores
Description: Chronic Pain Acceptance Questionnaire-Revised. Scores range from 0-120 with higher scores representing higher chronic pain acceptance, a better outcome.
Time Frame: Baseline and 4 weeks (pre to post-intervention)
Population: Participants who completed baseline and post assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training
Number analyzed (Participants) | 22
score on a scale
  Pre | 57.64 (4.22)
  Post | 70.91 (4.46)
Statistical Analysis 1: Comparison: Mindfulness Training; Test type: Other — Within-group paired t-test; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 13.27, 95% CI 2-sided [8.47 to 18.07], Standard Error of Mean 2.45

15. Other Pre Specified Outcome: Trait Mindfulness Scores
Description: Freiburg Mindfulness Inventory. Possible scores range from 14 to 52, with higher scores indicating greater mindfulness, a better outcome.
Time Frame: Baseline and 4 weeks (pre to post-intervention)
Population: Participants who completed baseline and post assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Training
Number analyzed (Participants) | 22
score on a scale
  Pre | 34.23 (12.79)
  Post | 42.23 (8.10)
Statistical Analysis 1: Comparison: Mindfulness Training; Test type: Other — Within-group paired t-test; p = 0.001, t-test, 2 sided; Mean Difference (Final Values) = 8.00, 95% CI 2-sided [3.92 to 12.08], Standard Error of Mean 1.96

ADVERSE EVENTS:
Time Frame: 4 weeks (session 1 through session 4)
Arm/Group | Mindfulness Training
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 1/23
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Training (N=23)
Distress due to potential for dissociating (Psychiatric disorders) | 1 (1) — Participant felt like might dissociate during mindfulness meditation practice (had past history of a dissociative disorder). Resulted in distress, which was resolved during the course of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT03495856/Prot_SAP_000.pdf